CLINICAL TRIAL: NCT07017231
Title: The Role of the Interleukin-13 Pathways on Pain and Itch Sensitivity in Patients With Atopic Dermatitis and Healthy Volunteers
Brief Title: Role of Interleukin-13 Pathways on Pain and Itch Sensitivity ( IL-13 )
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Silvia Lo Vecchio, Associate Professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20240029 2nd subproject
Record Dates: First submitted 2025-05-30; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Itching
MeSH Terms: conditions — Pruritus | interventions — Histamine

STUDY DESIGN:
Intervention Model Description: Each participant will be treated with Lebrikizumab and will receive 2 pruritogens:
  Histamine and cowhage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lebrikizumab (Experimental): The initial doses will be subcutaneous Lebrikizumab 500 mg (two 250 mg injections) at both week 0 (baseline) and week 2, followed by 250 mg administered subcutaneously at week 4.
  Interventions: Other: histamine dihydrochloride; Other: Cowhage

INTERVENTIONS:
Other: histamine dihydrochloride — A small drop of histamine dihydrochloride (1%, in saline) will be applied to two previously determined areas followed by a prick through the drop.
Other: Cowhage — Approximately 30-35 cowhage spicules will be manually inserted into the subject's skin.

SUMMARY:
Atopic dermatitis (AD) is as chronic, inflammatory skin disorder affecting 20% of the world's population. Intense itch and skin pain are the main symptoms. Research has shown that the proteins interleukins are involved in inflammation and itch in atopic dermatitis. The medicinal product called Lebrikizumab, used for treatment of AD, has shown to block the interleukin called IL-13. The purpose of this experiment is to evaluate the role of IL-13 in itch in people with atopic dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is as chronic, inflammatory skin disorder affecting 20% of the world's population. Intense itch and skin pain are the main symptoms. Research has shown that the interleukin-13 is involved in inflammation and itch in atopic dermatitis by increasing the neuronal sensitivity to pruritogens.

However, the physiological mechanisms by which IL-13 increases the itch sensitivity are unclear. The aim of this project is to use, for the first time in humans, the monoclonal antibody Lebrikizumab that inhibits IL-13 with high affinity as a novel experimental tool to modulate the IL-13 pathway and evaluate its role in the transmission and processing of itch and pain.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years • The patients should have an AD according to diagnosis by a board-certified dermatologist, with an Eczema Area and Severity Index (EASI), a validated scoring tool that grades the physical signs of AD of at least 7. The project team will be specifically trained and evaluated in the EASI assessment to ensure interindividual consistency.

Exclusion Criteria:

* Pregnancy or lactation

  * Drug addiction defined as any use of cannabis, opioids, or other drugs Moles, wounds, scars, or tattoos in the area to be treated or tested
  * Treatment within two weeks before start of the experiment with topical corticosteroids or calcineurin inhibitors.
  * Treatment within two weeks before start of the experiment with topical treatments (excluding emollients) on the skin areas selected for testing (eight weeks if treated with systemic treatments for AD such as methotrexate or azathioprine)
  * Treatment with antihistamines 72 hours before start of the experiment
  * Previous or current history of neurological, musculoskeletal, cardiac disorder, or psychiatric diagnoses that may affect the results (e.g., neuropathy, muscular pain in the upper extremities, anxiety, depression, schizophrenia, etc.)
  * Current use of medications that may affect the trial such as antihistamines and painkillers (use of antihistamines must be discontinued 72 hours before the experiment and all topical agents and emollients must be discontinued 24 hours before the experiment).
  * Use of systemic corticosteroids
  * Consumption of alcohol or painkillers 24 hours before the study days and between these
  * Participation in other trials within one week of study entry (four weeks in the case of pharmaceutical trials)
  * Lack of ability to cooperate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measuring itch by computerized Visual Analog Scale Scoring | Day 1
  The subjects will be asked to rate the sensation of itch on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no itch" and 100 indicates "worst itch imaginable".
Superficial blood perfusion | Day 1
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Wheal reaction | Day 1
  Wheal reaction measurement will be conducted immediately after the removal of pruritogens by measuring the longest diameter with a ruler.
Average pruritis and pain numerical rating scale (NRS) | Day 1
  The subject will be asked to retrospectively rate the average and worst itch/pain on an 11-point scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)experience they had during the last 7 days.
Skin peak pain numerical rating scale (SPP-NRS) | Day 1
  According to the SPP-NRS, the subject will be asked about "worst skin pain" they felt in the past 24 hours on an 11- point scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Peak pruritus numerical rating scale (PP-NRS) | Day 1
  The subject will be asked about the "worst itch" they felt in the past 24 hours on an 11-point scale ranging from 0 to 10 (0 = no itch and 10 = worst imaginable itch)
Eczema Area and Severity Index (EASI) | Day 1
  This scale is used for patients with AD to assess severity and extent of the disease. The investigator/physician will assign scores based on redness, scratching, thickness, lichenification and percentage of affected body regions
Dermatology Life Quality Index (DLQI) | Day 1
  This questionnaire is a simple 10-question validated questionnaire that measures the impact of the skin disease on several aspects of the patient's life over the past week. The DLQI sum score is calculated by summing up the score of each item. Questions are scored on a four-point Likert scale: 0, not at all/not relevant; 1, a little; 2, a lot; and 3, very much.
Itch Severity Scale (ISS) | Day 1
  This is a seven items questionnaire: itch description, frequency, effect on sleep, effect on mood, effect on sexual desire/function, itch intensity using Likert scale and body surface area involved
Patient Oriented Eczema Measure (POEM) | Day 1
  POEM is a questionnaire used for patients' self-monitoring of AD severity. It asks about the frequency of seven symptoms (itch, sleep disturbance, dryness, flaking, weeping, or oozing, bleeding, and cracking) in the past seven days, and the patient has to choose between these answers: No days, 1-2 days, 3-4 days, 5-6 days, Every day
Mechanically evoked itch (MEI) | Day 1
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Mechanically evoked itch (MEI) | Day 3
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).
Measuring pain by computerized Visual Analog Scale Scoring | Day 3
  The subjects will be asked to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Measuring pain by computerized Visual Analog Scale Scoring | Day 4
  The subjects will be asked to rate the sensation of pain on a 100 mm VAS scale ranging from 0 to 100 where 0 indicates "no pain" and 100 indicates "worst pain imaginable".
Superficial blood perfusion | Day 3
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Superficial blood perfusion | Day 4
  Superficial blood perfusion (SBP) is measured by a Speckle contrast imager
Wheal reaction | Day 3
  Wheal reaction measurement will be conducted immediately after the removal of pruritogens by measuring the longest diameter with a ruler.
Wheal reaction | Day 4
  Wheal reaction measurement will be conducted immediately after the removal of pruritogens by measuring the longest diameter with a ruler.
Average pruritis and pain numerical rating scale (NRS) | Day 3
  The subject will be asked to retrospectively rate the average and worst itch/pain on an 11-point scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)experience they had during the last 7 days.
Average pruritis and pain numerical rating scale (NRS) | Day 4
  The subject will be asked to retrospectively rate the average and worst itch/pain on an 11-point scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)experience they had during the last 7 days.
Skin peak pain numerical rating scale (SPP-NRS) | Day 3
  According to the SPP-NRS, the subject will be asked about "worst skin pain" they felt in the past 24 hours on an 11- point scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Skin peak pain numerical rating scale (SPP-NRS) | Day 4
  According to the SPP-NRS, the subject will be asked about "worst skin pain" they felt in the past 24 hours on an 11- point scale ranging from 0 to 10 (0 = no pain and 10 = worst imaginable pain)
Peak pruritus numerical rating scale (PP-NRS) | Day 3
  The subject will be asked about the "worst itch" they felt in the past 24 hours on an 11-point scale ranging from 0 to 10 (0 = no itch and 10 = worst imaginable itch)
Peak pruritus numerical rating scale (PP-NRS) | Day 4
  The subject will be asked about the "worst itch" they felt in the past 24 hours on an 11-point scale ranging from 0 to 10 (0 = no itch and 10 = worst imaginable itch)
Eczema Area and Severity Index (EASI) | Day 3
  This scale is used for patients with AD to assess severity and extent of the disease. The investigator/physician will assign scores based on redness, scratching, thickness, lichenification and percentage of affected body regions
Eczema Area and Severity Index (EASI) | Day 4
  This scale is used for patients with AD to assess severity and extent of the disease. The investigator/physician will assign scores based on redness, scratching, thickness, lichenification and percentage of affected body regions
Dermatology Life Quality Index (DLQI) | Day 3
  This questionnaire is a simple 10-question validated questionnaire that measures the impact of the skin disease on several aspects of the patient's life over the past week. The DLQI sum score is calculated by summing up the score of each item. Questions are scored on a four-point Likert scale: 0, not at all/not relevant; 1, a little; 2, a lot; and 3, very much.
Dermatology Life Quality Index (DLQI) | Day 4
  This questionnaire is a simple 10-question validated questionnaire that measures the impact of the skin disease on several aspects of the patient's life over the past week. The DLQI sum score is calculated by summing up the score of each item. Questions are scored on a four-point Likert scale: 0, not at all/not relevant; 1, a little; 2, a lot; and 3, very much.
Itch Severity Scale (ISS) | Day 3
  This is a seven items questionnaire: itch description, frequency, effect on sleep, effect on mood, effect on sexual desire/function, itch intensity using Likert scale and body surface area involved
Itch Severity Scale (ISS) | Day 4
  This is a seven items questionnaire: itch description, frequency, effect on sleep, effect on mood, effect on sexual desire/function, itch intensity using Likert scale and body surface area involved
Patient Oriented Eczema Measure (POEM) | Day 3
  POEM is a questionnaire used for patients' self-monitoring of AD severity. It asks about the frequency of seven symptoms (itch, sleep disturbance, dryness, flaking, weeping, or oozing, bleeding, and cracking) in the past seven days, and the patient has to choose between these answers: No days, 1-2 days, 3-4 days, 5-6 days, Every day
Patient Oriented Eczema Measure (POEM) | Day 4
  POEM is a questionnaire used for patients' self-monitoring of AD severity. It asks about the frequency of seven symptoms (itch, sleep disturbance, dryness, flaking, weeping, or oozing, bleeding, and cracking) in the past seven days, and the patient has to choose between these answers: No days, 1-2 days, 3-4 days, 5-6 days, Every day
Mechanically evoked itch (MEI) | Day 4
  MEI is measured by using mildly pruritic, non-painful von Frey nylon filaments of a predetermined intensity (generally 5-30 miliNewton of force).

SECONDARY OUTCOMES:
Mechanical Pain Thresholds (MPT) | Day 1
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Sensitivity (MPS) | Day 1
  This test is conducted with the same pinprick set used to test the MPT.
Pressure Pain Thresholds (PPT) | Day 1
  Pressure will be applied by a handheld electronic pressure algometer (Somedic AB, Stockholm, Sweden) on to the supinator muscle on the left forearm.
Cold Detection Thresholds (CDT) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Day 1
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Mechanical Pain Thresholds (MPT) | Day 3
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Thresholds (MPT) | Day 4
  This test is conducted using a pinprick set. The set consists of 7 needles each with a diameter of 0.6 mm and different force applications: 8, 16, 32, 64, 128, 256, and 512 mN.
Mechanical Pain Sensitivity (MPS) | Day 3
  This test is conducted with the same pinprick set used to test the MPT.
Mechanical Pain Sensitivity (MPS) | Day 4
  This test is conducted with the same pinprick set used to test the MPT.
Pressure Pain Thresholds (PPT) | Day 3
  Pressure will be applied by a handheld electronic pressure algometer (Somedic AB, Stockholm, Sweden) on to the supinator muscle on the left forearm.
Pressure Pain Thresholds (PPT) | Day 4
  Pressure will be applied by a handheld electronic pressure algometer (Somedic AB, Stockholm, Sweden) on to the supinator muscle on the left forearm.
Cold Detection Thresholds (CDT) | Day 3
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thrteshold | Day 1
Cold Detection Thresholds (CDT) | Day 4
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Day 3
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Warm Detection Thresholds (WDT) | Day 4
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Heat Pain Thrteshold | Day 3
Heat Pain Thrteshold | Day 4
Pain to Supra-threshold Heat Stimuli (STHS) | Day 4
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Day 3
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Cold Pain Thresholds (CPT) | Day 4
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device
Pain to Supra-threshold Heat Stimuli (STHS) | Day 3
  The tests of thermal sensation will all be conducted using a TSA2 (Medoc Ltd, Israel) thermal sensory testing device

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Neuroplasticity and Pain Faculty of Medicine, Aalborg University Selma Lagerløfs Vej 249 9260 Gistrup, Denmark, Gistrup, Denmark